CLINICAL TRIAL: NCT01887847
Title: A Randomized, 2 Way Crossover, Pilot Pharmacokinetic Study of Investigational Sublingual Nicotine Tablets ( Pharmaceutical Productions Inc.) Versus COMMIT Smoking Lozenge ( GLAXOSMITHKLINE) in Healthy Smoking Volunteers
Brief Title: Pilot Pharmacokinetic Study of Investigational Sublingual Nicotine Tablet Versus COMMIT Nicotine Lozenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Productions Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PPI 2006-01; R41DA033710 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-27 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Nicotine Pharmacokinetic Study
Keywords: nicotine; pharmacokinetics
MeSH Terms: interventions — Nicotine; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sublingual nicotine tablet (Experimental): investigational 2 mg sublingual nicotine tablet
  Interventions: Drug: Nicotine (Pharmaceutical Productions Inc.)
- COMMIT nicotine lozenge (Active Comparator): COMMIT 2 mg nicotine lozenge
  Interventions: Drug: Nicotine (Pharmaceutical Productions Inc.)

INTERVENTIONS:
Drug: Nicotine (Pharmaceutical Productions Inc.) — An investigational 2 mg sublingual nicotine tablet (Pharmaceutical Productions Inc.) will be administered in a randomized crossover design in 6 male and female otherwise healthy smokers.
  Other Names: Investigational 2 mg sublingual nicotine tablet
  Arms: sublingual nicotine tablet
Drug: Nicotine (Pharmaceutical Productions Inc.) — A Commit® 2 mg nicotine lozenge (GlaxoSmith Kline)will be administered in a randomized crossover design in 6 male and female otherwise healthy smokers.
  Other Names: Commit® 2mg nicotine lozenge (GlaxoSmith Kline)
  Arms: COMMIT nicotine lozenge

SUMMARY:
The objective of this study is to compare the pharmacokinetics of an investigational 2 mg sublingual nicotine tablet (Pharmaceutical Productions Inc.) to a 2 mg Commit® nicotine lozenge (GlaxoSmith Kline) in a randomized crossover design in 6 male and female otherwise healthy smokers.

DETAILED DESCRIPTION:
A single oral dose of each medication will be administered to each participant with a 48 hour washout period between administrations. Serial blood samples will be obtained at the following times after the administration of the nicotine dosage forms: 0, 4, 8, 10, 12, 16, 30, 45, 60, 90, 120, and 180 minutes. Vital signs will be obtained prior to dosing and at 30, 60, 180, and 240 minutes after dosage administration. A craving questionnaire will be administered prior to dosing and at 5, 11, 17, 25, 35, 50, and 65 minutes. Craving questionnaires will then be administered at 30 minute intervals thereafter up to 180 minutes after medication administration. A Product Preference Questionnaire will be completed at the end of the second study period. A 30 day follow-up visit will be scheduled with each participant at the conclusion of the study

ELIGIBILITY:
Inclusion Criteria:

* Subjects have to be 18-45 years old
* Subjects must provide written informed consent prior to any study related procedures being performed.
* Subjects must have a willingness and ability to comply with the protocol requirements.
* Subjects must be in good health and free from any clinically significant pathology (gastrointestinal tract, hepatic, renal, cardiovascular, central nervous system diseases)
* Subjects must have body mass index not to exceed 35
* Female subjects of childbearing potential, in addition to having a negative urine pregnancy test, must be willing to use a form of birth control during the study. The hormonal contraceptives should be avoided within 2 month prior to study entry.
* Subjects must consume more than 15 cigarettes daily and smoke their first cigarette within 30 minutes of awaking from sleeping.
* A Fagerstrom Smoking index greater than 4

Exclusion Criteria:

* Subjects that have used other nicotine delivery system such as nicotine lozenge, nicotine patch, nicotine inhaler, or nicotine nasal spray etc. within 30 days of study entry.
* Subjects who have smoked any substance other than tobacco within 30 days of study entry.
* Subjects that have used other smoking cessation aids (including bupropion, herbals, counseling, etc.) within 30 days of study entry.
* Subjects who have currently involved in another clinical trial or have used any investigational drug within 3 month of study entry.
* Subject who is pregnant or lactating, or planned to became pregnant within 6 months.
* Subjects who have diagnosed heart disease or are being treated with medication or had an irregular heartbeat or have had a heart attack.
* Subject with diagnosed stomach ulcers.
* Subjects who have taking insulin for diabetes.
* Subjects with high blood pressure not controlled by medication or a blood pressure greater than 150 mmHg systolic or 90 mmHg diastolic
* Subjects who are unable to fulfill study requirements in relation to conforming to the visit schedule.
* Subjects who have severe allergic history
* Subjects who have known intolerance to medication
* Subjects who have diagnosed chronic diseases of cardiovascular, pulmonary, neuro-endocrine systems, gastrointestinal, hepatic, renal, and blood diseases
* Subjects who had surgical operations on gastrointestinal tract with the exception of appendectomy
* Subjects who had acute infectious diseases within the last 4 weeks prior to the study entry;
* Subjects who donated 450 mL and more of his/her blood or blood plasma within the last 2 month prior to the study entry
* Subjects who are taking more than 10 units of alcohol per week or have a history of alcohol and drug abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is to substantiate that the pharmacokinetics of this novel nicotine replacement therapy (NRT) resembles that of smoking a cigarette, wherein the average Tmax is about 15 minutes or less. ► | Serial blood samples will be obtained at the following times after the administration of the nicotine dosage forms: 0, 4, 8, 10, 12, 16, 30, 45, 60, 90, 120, and 180 minutes.

SECONDARY OUTCOMES:
The secondary outcome is to compare craving scores for this investigational nicotine replacement therapy (NRT) to the lozenge. | A craving questionnaire will be administered prior to dosing and at 5, 11, 17, 25, 35, 50, and 65 minutes and will then be administered every 30 minute thereafter up to 180 minute.
  A craving questionnaire will be administered prior to dosing and at 5, 11, 17, 25, 35, 50, and 65 minutes. Craving questionnaires will then be administered at 30 minute intervals thereafter up to 180 minutes after medication administration.
A Product Preference Questionnaire | At the end of the second dosing day.
  At the end of the second dosing day the participant will be asked to fill out the Patient Preference Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vocci, Ph.D, Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute Clinic, Torrance, California, United States